CLINICAL TRIAL: NCT02479464
Title: A Pilot Study for the Evaluation of the Clinical Impact of the Antidepressant Pharmacogenomic Algorithm in an Outpatient Therapy-based Clinical Setting
Brief Title: Clinical Impact of the Antidepressant Pharmacogenomic Algorithm in an Outpatient Therapy-based Clinical Setting
Acronym: HAMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: AssureRx Health, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel K. Hall-Flavin, Associate Professor of Psychiatry, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09-002523
Record Dates: First submitted 2015-06-16; First posted 2015-06-24 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
Keywords: AssureRx; Algorithm; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (No Intervention): This is the treatment as usual arm to monitor the current standard clinical practice
- Part 2 (Other): This group will be provided with genotyping results after baseline visit to guide clinical medication management
  Interventions: Genetic: Genotyping results

INTERVENTIONS:
Genetic: Genotyping results — Genotyping results provided in Phase II
  Arms: Part 2

SUMMARY:
The Mayo Clinic psychiatric pharmacogenomic team has developed a pharmacogenomic algorithm that has been designed to improve the effectiveness and safety of antidepressant medications by providing guidance in medication selection and appropriate dosing. This algorithm has been incorporated into a new genotyping interpretative report. This report is now available from AssureRx. The pharmacogenomic algorithm is based on genotyping both copies of four informative genes. These four genes are: 1) the Cytochrome P450 2D6 gene; 2) the Cytochrome P450 2C19 gene; 3) the Serotonin Transporter gene (SLC6A4); and 4) the Serotonin 2A receptor gene (5HTR2A). Though this algorithm is not yet part of the universal standard of care, Mayo clinicians have found it helpful in guiding treatment decisions at Mayo Clinic Rochester.

DETAILED DESCRIPTION:
The proposed pilot study is designed to evaluate the clinical impact of the interpretive report in an outpatient behavioral health clinic in St. Paul, Minnesota. While the ultimate goal of this project is to show an improvement in patient outcomes, this pilot study will be used to evaluate the feasibility of introducing the pharmacogenomic algorithm to a new setting that does not routinely use the algorithm. Secondary outcome data will be collected to generate meaningful estimates of the magnitude of potential treatment effects. The study will consist of two phases, each enrolling 2530 subjects. In Phase 1, consecutive patients will be prospectively monitored to observe standard practice. Patients will be given the option to receive genotyping and those that agree will have blood drawn. However, the results of the genotyping and algorithm will not be released until all phase 1 patients have completed study visits.. Subsequently, in Phase 2, also enrolling 3025 subjects, the results of the genotyping and algorithm will be made available immediately for additional consecutive prospectively monitored patients. Patients will be prospectively monitored in the same fashion as Phase 1. The results of the study will be used to perform preliminary analyses and subsequent fully powered multi-site trials will be planned based on the results of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between the ages of 18 and 80.
2. Major depressive disorder or depressive disorder not otherwise specified (NOS) as ascertained by a physician or mental health professional licensed to diagnose.
3. Patient is an outpatient and not in imminent need of inpatient hospitalization
4. Patient's Hamilton Depression Rating score is >14
5. Patient is being seen by a psychiatrist for optimum medication management.
6. Ability to read, understand and sign an informed consent document

Exclusion Criteria:

1. Serious medical illness (as ascertained via the initial triage screening process)
2. Patients with a diagnosis of Bipolar I disorder
3. Patients with a diagnosis of Schizophrenia or Schizoaffective disorder
4. Patients who are legally unable to consent to enrollment in the study (i.e. patients with legal guardians)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients approached who consent to use of pharmacogenomic algorithm | 8 weeks
Amount of time from ordering test to receipt of results | 8 weeks
Proportion of time that the physician prescribed a medication that was recommended by the algorithm | 8 weeks

SECONDARY OUTCOMES:
Time to remission of depressive symptoms | 8 weeks
  Hamilton rating of < 7
Measured side effect burden | 8 weeks
  Reduction in Frequency, Intensity, and Burden of Side Effects Rating (FIBSER) score.
Number of participants who change their initial medication regimen | 8 weeks
Health care clinical cost | 8 weeks
  defined by analysis of mental health resource utilization
Physician satisfaction with delivery of clinical care | 8 weeks
  defined by researcher developed Likert-based satisfaction survey
Patient satisfaction with clinical care | 8 weeks
  defined by researcher developed Likert-based satisfaction survey

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials